CLINICAL TRIAL: NCT04879134
Title: Apomorphine Effect on Pain in Parkinson's Disease: A Randomized, Double-blind Placebo Cross-over Study
Brief Title: Apomorphine Effects on Pain in Parkinson's Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Paladin Labs Inc. (Other)
Responsible Party: Principal Investigator, Veronica Bruno, Clinical Assistant Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: REB20-0423
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: We will perform a small pilot double-blind, randomized cross-over study evaluating the safety and efficacy of apomorphine injections vs. placebo injections on pain in PD. Subjects, caregivers, and investigators will be blinded to the assignment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Upon entry to the study, all subjects will be assigned to a subject number. Eligible subjects will be randomized to receive either apomorphine injections or placebo on VISIT 2 in a double-blind manner according to a randomization schedule using computerized randomization tables prepared by a blinded clinical nurse. Participants will then cross over to the other treatment group to receive apomorphine or placebo injections on VISIT 3. The specific type of randomization used will be block randomization to ensure equal sample sizes of the apomorphine and placebo groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apomorphine Injections (Experimental)
  Interventions: Drug: Apomorphine Injectable Solution
- Placebo Injections (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apomorphine Injectable Solution — Patients will receive the treatment while they are in an OFF period, without the effect of any antiparkinsonian medication. For this study, the initial dose of apomorphine or placebo will be 2 mg. We selected an initial standardized dose based on the pharmacological characteristics of apomorphine. Assessments will be completed 30 and 60 minutes after the initial dose. At 60 minutes from the first dose, a 3 mg dose will be administered, and again, assessments will be completed after 30 and 60 minutes. The total given dosage will be 5 mg. Blood pressure and pulse will be checked every 20 minutes after injections.
  Other Names:
  Movapo
  Arms: Apomorphine Injections
Drug: Placebo — 0.9% saline placebo injection
  Other Names:
  • Saline
  Arms: Placebo Injections

SUMMARY:
To study the effects of acute apomorphine vs. placebo administration on different Parkinson's disease pain types.

DETAILED DESCRIPTION:
Apomorphine is the only anti-parkinsonian agent compatible with levodopa in improving Parkinson's disease (PD) motor symptoms. Besides, it has positive effects on some of the nonmotor symptoms of the disease, such as urinary disturbances and sleep. Apomorphine is usually well tolerated as it produces limited side effects. Knowledge about the effects of apomorphine on pain in PD is scarce. Evidence on this topic has only been reported in case reports or small studies but represents a potentially important use of the drug. We hypothesize that apomorphine may be a rational, safe, and useful treatment for subjects with pain in PD, including different subtypes. Within this framework, the present study will evaluate the effect of acute apomorphine vs. placebo administration on different PD pain types.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with PD according to the MDS Clinical diagnostic criteria for Parkinson's disease.
* Participants on antiparkinsonian medication in advanced stages of the disease and experiencing OFF periods and pain.
* Apomorphine treatment naïve subjects or not received any within the last six months.
* Stable PD and pain medications for at least 30 days.
* Competence to self-report pain severity in the King's Parkinson's disease Pain Scale and a Likert Visual Analogue Scale.

Exclusion Criteria:

* Subjects who are unable to self-report pain severity in the selected scales. Patients that may require a translator or are illiterate will be included if they can self-report pain severity.
* Subjects with a diagnosis of dementia (Montreal Cognitive Assessment <20).
* Subject with poorly controlled orthostatic hypotension.
* Subjects associated with another medical condition, e.g., any cardiovascular, renal or hepatic impairment, hematological or psychiatric diseases.

Any contraindication to receiving apomorphine injections:

* Subjects who are hypersensitive to apomorphine or any ingredient in the formulation or component of the container (hydrochloric acid concentrated, sodium bisulfite (E222), and water)
* Subjects using concomitant drugs of the 5HT3 antagonist class including (e.g., ondansetron, granisetron, palonosetron)
* Subjects using concomitant antihypertensive medications or vasodilators
* Subjects with prolonged QT on an electrocardiogram.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Unified Parkinson Disease Rating Scale | 0, 1 and 2 weeks
  Measures changes of symptom severity, treatment response and the efficacy of treatments. Part 1 (non-motor experiences of daily living), Part 2 (motor experiences of daily living), Part 3 (motor examination) and Part 4 (motor complications). The maximum score for all the parts is 272. Higher scores are indicative of worse outcomes.
Change in Likert Visual Analogue Scale | 0, 1 and 2 weeks
  The measure of global pain change perceived by the patients. The most simple Likert Visual Analogue Scale is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom, pain, health) orientated from the left (worst) to the right (best). There are no numerical values on this scale however, a positioning towards the left of the scale indicates a worse outcome.

SECONDARY OUTCOMES:
Change in Clinical Global Impression Scale | 0, 1 and 2 weeks
  Changes in scores on the Clinical Global Impression (CGI) scale. CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).CGI scores range from 1 (very much improved) through to 7 (very much worse). Treatment response ratings should take account of both therapeutic efficacy and treatment-related adverse events and range from 0 (marked improvement and no side-effects) and 4 (unchanged or worse and side-effects outweigh the therapeutic effects). Each component of the CGI is rated separately; the instrument does not yield a global score.
Number of adverse events | 0, 1 and 2 weeks
  Adverse events assessed for safety purposes at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Bruno, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- Movement Disorder Program, Foothills Medical Center, Alberta Health Services, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No